CLINICAL TRIAL: NCT03237559
Title: A Descriptive Comparative Study to Assess Knowledge, Attitude and Practice Regarding Eugenics Among Eligible Couples of Selected Area of Ambala, Haryana (India)
Brief Title: Assessment of Knowledge, Attitude and Practice of Eligible Couples Regarding Eugenics
Status: Completed | Type: Observational
Sponsor: Maharishi Markendeswar University (Deemed to be University) (Other)
Responsible Party: Principal Investigator, Hem Sadhanu, Student M.Sc.Nursing, Maharishi Markendeswar University (Deemed to be University)
Other Study IDs: 781
Record Dates: First submitted 2017-07-30; First posted 2017-08-02 (Actual); Last update posted 2017-08-02 (Actual); Status verified 2017-07

CONDITIONS: Knowledge, Attitudes, Practice
Keywords: Eugenics; Eligible Couples; Knowledge; Attitude; Practice
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- eligible couples: Eligible couples refers to methods that are adopted by eligible couples for having physically and psychologically healthy conception and pregnancy

SUMMARY:
A Descriptive study to assess the knowledge, attitude and practice regarding eugenics among eligible couples of selected area of Ambala, Haryana, India. Eligible couples were the married couples where wife is in the age group of 15-45 years planning for conception, have conceived and may or may not have any living child.Eugenics are to methods that are adopted by eligible couples for having physically and psychologically healthy conception and pregnancy.

DETAILED DESCRIPTION:
To assess the knowledge, attitude and practice the structured knowledge questionnaire, attitude 5-point likert scale and expressed checklist tool were prepared. A sample size of 318 was calculated by power analysis and eligible couples were selected by Purposive sampling technique from rural and urban area of Ambala Haryana, India.

Each eligible couples (separately husband and wife) data was collected through Self- Report technique.one time assessment only done.

ELIGIBILITY:
Inclusion Criteria:

* who were present at the time of data collection
* who were willing to participate in the study
* who can read and write English/Hindi

Exclusion Criteria:

* who have more than 2 children
* who had undergone permanent sterilization

Ages: 15 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Wife
Study Population: Eligible couples of rural and urban areas of Ambala Haryana, India
Sampling Method: Non-Probability Sample
Enrollment: 318 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Structured Questionnaire | 15-20 min
  It consisted of 34 knowledge items to assess the knowledge of Eligible couples regarding Eugenics. The following content areas were:
  * Concept of Eugenics
  * Screening of Disease
  * Nutrition
  * Vaccination
  * Lifestyle
  * Exposure to substance abuse or toxins All 34 test items were multiple choice questions. Each item had a single correct answer. Every correct answer was awarded a score of '1' and every incorrect answer was assigned a score of 00. The maximum possible score was 34 and minimum score was 00 on the structured knowledge questionnaire . Higher score indicated that eligible couples have good knowledge regarding Eugenics. Based on scoring criteria on Structured Knowledge Questionnaire, knowledge was categorized into four level of knowledge.Excellent (27-34),Good (21-26),Average (17-20),Below average(0-16)

SECONDARY OUTCOMES:
Structured Attitude 5-point likert Scale | 10-15 min
  Scale consisted of 30 items on which the respondent had to respond on 5- points Likert's scale.Each statement score was divided as strongly agree, agree, undecided, disagree, strongly disagree (maximum score was 150 and minimum score was 30).Tool had 15 positive items and 15 negative items.Positive statements were scored SA (Strongly Agree) -5, A (Agree)-4, U (Undecided)-3, D (Disagree)-2, SD (Strongly Disagree)-1. Negative statements were scored SA (Strongly Agree) -1, A (Agree)-2, U (Undecided)-3, D (Disagree)-4, SD (Strongly Disagree)-5.
  Based on scoring criteria on Structured Attitude Scale, Husbands and Wives attitude was categorized into three level of Attitude Favourable (225-300), Moderately Favourable(180-224),Unfavourable(60-179)
Expressed Husband Checklist | 7-8min
  Structured expressed practice checklist was developed to assess expressed practices of Husbands regarding Eugenics. Checklist consists of 18 items. These items designed to elicit information on practices of Husbands regarding Traditional and Non-traditional. Each item was provided with 2 responses Yes(Y) and No (N) and was scored as 1 and 0 respectively.
Expressed Wife Checklist | 10-12min
  Structured expressed practice checklist was developed to assess expressed practices of wives regarding Eugenics. Checklist consists of 32 items. These items designed to elicit information on practices of wives regarding Traditional and Non-traditional. Each item was provided with two responses Yes(Y) and No (N) and was scored as 1 and 0 respectively

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Poonam Sheoran, Ph.d Nursing, Study Director — M.M.University, Mullana, Ambala Haryana, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Okka B, Durduran Y, Degerli Kodaz N. Traditional practices of Konya women during pregnancy, birth, the postpartumperiod, and newborn care. Turk J Med Sci. 2016 Feb 17;46(2):501-11. doi: 10.3906/sag-1504-120. PMID 27511518
- [Background] Charafeddine L, El Rafei R, Azizi S, Sinno D, Alamiddine K, Howson CP, Walani SR, Ammar W, Nassar A, Yunis K. Improving awareness of preconception health among adolescents: experience of a school-based intervention in Lebanon. BMC Public Health. 2014 Jul 31;14:774. doi: 10.1186/1471-2458-14-774. PMID 25081733